CLINICAL TRIAL: NCT05130359
Title: Explore Whether Banana Peel Extract Can Improve Sleep
Brief Title: Evaluation of the Sleep-relieving Effect of Banana Peel Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202103033
Record Dates: First submitted 2021-10-21; First posted 2021-11-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Impaired Attention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): take 2 tablets 2 hours before bedtime for 4 consecutive weeks
  Interventions: Dietary Supplement: Placebo
- Banana peel extract (Experimental): take 2 tablets 2 hours before bedtime for 4 consecutive weeks
  Interventions: Dietary Supplement: Banana peel extract

INTERVENTIONS:
Dietary Supplement: Placebo — take 2 tablets 2 hours before bedtime for 4 consecutive weeks
  Arms: Placebo
Dietary Supplement: Banana peel extract — take 2 tablets 2 hours before bedtime for 4 consecutive weeks
  Other Names: Happy Banana
  Arms: Banana peel extract

SUMMARY:
Banana peel has the potential to improve sleep quality. The purpose of this research is to test the effect of banana peel on improving sleep quality.

DETAILED DESCRIPTION:
Insomnia is one of the most frequently complained sleep problems in sleep disorders, and in recent years has been regarded by the medical community as a disease that seriously affects people's lives and quality of life. The problem of perishable and perishable causes a great burden on the environment. However, banana peels actually contain many functional ingredients, such as dietary fiber, minerals, alkaloids, flavonoids, phenols, saponins, tannins and dopamine, etc. Banana peel contains more total phenols and total flavonoids than banana pulp. Studies have pointed out that banana peel extraction can inhibit the growth of fungi and bacteria. In addition, it also has antioxidant, anti-depressant, and diuretic functions. Banana peel can also improve the performance of tryptophan metabolism-related genes

ELIGIBILITY:
Inclusion Criteria:

1.20 to 65-year-old males or non-pregnant females who are willing to sign the subject's consent.

2.Pittsburgh Sleep Quality Index (PSQI) score> 5

Exclusion Criteria:

1. Taking sleeping pills and melatonin
2. People suffering from mental illness
3. Pregnant or breastfeeding women
4. People who are known to be allergic to bananas
5. Have heart-related diseases
6. People with symptoms of sleep cessation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Sleep monitoring | at 4 week after taking test sample
  Detect the electrical activity of the heart in the potential difference between two specific points on the body surface to reflect the state of sleep
Serotonin | at 4 week after taking test sample
  Venous blood was sampled to measure concentrations of Serotonin
Melatonin | at 4 week after taking test sample
  Collect saliva samples in the morning upon waking to measure melatonin concentration.
Sleeping quality | at 4 week after taking test sample
  The Pittsburgh Sleep Quality Index (PSQI) will be utilized to assess sleeping quality. The minimum value is 0, the maximum value is 42. The higher the score, the worse the outcome.
Insomnia Severity | at 4 week after taking test sample
  The Insomnia Severity Index (ISI) will be utilized to assess insomnia severity. The minimum value is 0, the maximum value is 28. The higher the score, the worse the outcome.

OTHER OUTCOMES:
The change of liver function biomarkers (AST, ALT) of blood | at 4 week after taking test sample
  Fasting venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | at 4 week after taking test sample
  Fasting venous blood was sampled to measure renal function biomarkers
The change of fasting blood glucose | at 4 week after taking test sample
  Fasting venous blood was sampled to measure concentrations of blood glucose
The change of Blood lipids profiles (Total-Cholesterol, HDL-C, LDL-C, triglycerides) | at 4 week after taking test sample
  Fasting venous blood was sampled to measure concentrations of Blood lipids profiles (Total-Cholesterol, HDL-C, LDL-C, triglycerides)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Chien Lee, Doctor, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No